CLINICAL TRIAL: NCT06882187
Title: Outcomes of Acute Limb Ischemia in Cancer Patients .
Brief Title: ALI in Cancer Patients
Acronym: ALI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Sayed Ahmed Ahmed Morsy, Resident ., Assiut University
Other Study IDs: ALI in Cancer Patients .
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Acute Limb Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to describe and evaluate the outcomes of cancer patients presenting with and treated for ALI at our center .

DETAILED DESCRIPTION:
Acute limb ischemia (ALI) is a vascular emergency and is associated with significant morbidity and mortality. Peripheral arterial embolism or thrombosis from malignant disease is uncommon and a rare cause of acute limb ischemia. Limb ischemia can be caused by emboli from the tumor itself, from metastatic deposits within large vessels, as well as the tumors of adjacent organs such as the lung, which invade the left or right atrium of the heart and then disseminate to the main arteries of the body. This acute event may be the first indication of malignant disease in the patient.

ELIGIBILITY:
Inclusion Criteria:

* All cancer patient presented to Vascular and Endovascular surgery departement with ALI.

Exclusion Criteria:

* Patients with benign tumors or without active malignancy.
* Patients with iatrogenic limb ischemia related to a tumor chemoembolization procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients .
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Limb Salvage | baseline